CLINICAL TRIAL: NCT03194724
Title: Using Stable Isotope Techniques to Monitor & Assess the Vitamin A Status of Children Susceptible to Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Food Technology Research Centre, Botswana (Other Government)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); UNICEF (Other); University of Botswana (Other)
Responsible Party: Sponsor
Other Study IDs: RAF 6047
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Assessment of Vitamin A Status of Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Vitamin A exposure: There was no intervention
  Interventions: Other: Vitamin A supplementation
- Low vitamin A exposure: No intervention
  Interventions: Other: Vitamin A supplementation

INTERVENTIONS:
Other: Vitamin A supplementation — Bi annual vitamin A supplementation programme

SUMMARY:
The relationship between infections and malnutrition is synergistic, each further compromising the outcome of the other. Malnutrition compromises natural immunity leading to increased susceptibility to infections, more frequent and prolonged disease episodes, and increased severity of disease. Likewise, infections can aggravate or precipitate malnutrition through decreased appetite and food intake, nutrient malabsorption, nutrient loss or increased metabolic needs. Severe malnutrition often masks symptoms and signs of infectious diseases making prompt clinical diagnosis and treatment very difficult. Another issue is that infections (as well as overweight and obesity status) affect nutritional biomarkers making it difficult to assess the real magnitude of some nutritional problems. This is the case of vitamin A. Vitamin A deficiency is defined to be of severe public health importance if 20% or more of a defined population has a serum retinol concentration of less than 0.7 µmol/L.

DETAILED DESCRIPTION:
Vitamin A is an essential nutrient needed for the visual system, and maintenance of cell function for growth, epithelial integrity, red blood cell production, immunity and reproduction. All infants are born with low stores and depend on vitamin A from breast milk to initially accumulate and maintain adequate stores. Infants of vitamin A depleted women are at greater risk of becoming vitamin A deficient early in life, especially if they are not breast fed. Correcting vitamin A deficiency is addressed by some African countries through vitamin A supplementation of children and food fortification programs. However, assessing vitamin A status, and the effectiveness of government interventions, is challenging in settings where infectious diseases are endemic, as in most African countries. Evaluation of vitamin A status is relatively insensitive when based on changes in serum retinol concentrations, which are homeostatically controlled and negatively affected by subclinical infections. Liver stores of vitamin A, the best indicator of vitamin A status, cannot be routinely evaluated. The isotope dilution technique is the preferred method for determining vitamin A status and assessing the efficacy and effectiveness of intervention programs aimed at improving vitamin A status. It is the only indirect assessment method that provides a quantitative estimate of vitamin A status across the continuum of deficient to excessive stores. Thus, this technique can be used for assessing vitamin A status in populations at risk of excessive status due to exposure to too much vitamin A through combined supplementation and consumption of fortified foods and/or preformed vitamin A-rich foods. The aim of this project is to use nuclear techniques to evaluate vitamin A nutritional status of young children during semi-annual administration of vitamin A supplements, and to assess how this relates to infection status. The IAEA has provided significant support on use of stable isotopes in assessing body composition and breast milk to Member States in Africa, it is now establishing the stable isotope technique to assess vitamin A body stores in Cameroon and Zambia (and additional implementation is possible in Morocco) for use throughout the region. These inputs will be used in this project to provide key information to stakeholders on how vitamin A intervention programs affect vitamin A status in children and how infections affect vitamin A status or validity of stable isotope techniques.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included if they are in the target age range (3-5 years), are not planning to move from the study area for the duration of the study, and do not have severe illness at the time of enrolment

Exclusion Criteria:

* Exclusion criteria will generally include the following conditions: severe anaemia, severe acute malnutrition, obesity, or clinically defined severe illness, such as dehydration, severe diarrhoea or severe respiratory illness.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The project will include preschool children 3-5 years of age. This age has been selected given the high risk of vitamin A deficiency in young children, as well as national policy for biannual vitamin A supplementation of preschool children. Children younger than 3 will not be included due to the volume of blood needed for biomarker analysis. Recruitment will be done in various settings, including household-level, clinics/hospitals, and childcare centres.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-04-30 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Cross sectional vitamin A status | 1 year
  Vitamin A status determination using stable isotopes

SECONDARY OUTCOMES:
Assessment of the presence of clinical infections | 1 year
  Infections

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared for pooling purposes as this study is part of a regional project